CLINICAL TRIAL: NCT02215954
Title: A Phase III, Randomized, Assessor-Blinded, Parallel-Group, Multi-Centre, Clinical Study With FE 999169 for Oral Administration Versus Niflec® for Colon Cleansing: J-CLEAR
Brief Title: A Phase III Study With FE 999169 Versus Niflec for Colon Cleansing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 000176
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-04

CONDITIONS: Colon Cleansing in Preparation for Colonoscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment arm [1]: FE 999169 (Experimental): One sachet on the day before colonoscopy, and another sachet on the day of colonoscopy
  Interventions: Drug: FE 999169
- Treatment arm [2]: FE 999169 (Experimental): Two sachets on the day before colonoscopy
  Interventions: Drug: FE 999169
- Treatment arm [3]: Niflec (Active Comparator): One to two pack(s) on the day of colonoscopy
  Interventions: Drug: Niflec

INTERVENTIONS:
Drug: FE 999169 — FE 999169 is a white crystalline powder for oral solution. Each sachet (16.1 g) contains sodium picosulfate hydrate 10 mg, magnesium oxide 3.5 g and anhydrous citric acid 12 g as well as orange flavour, potassium bicarbonate and sodium saccharin as excipients. FE 999916 is dissolved by mixing the contents of the sachet with approximately 150mL of cold water in a cup before administration.
  Arms: Treatment arm [1]: FE 999169; Treatment arm [2]: FE 999169
Drug: Niflec — Niflec is a white-yellowish powder for oral solution. Each plastic sachet (137.155 g) contains sodium chloride 2.93 g, potassium chloride 1.485 g, sodium bicarbonate 3.37 g and sodium sulfate anhydrous 11.37 g, as well as macrogol 4000, saccharin sodium hydrate, flavour as excipients. Niflec is dissolved in water to make approximately 2 L of solution before administration.
  Arms: Treatment arm [3]: Niflec

SUMMARY:
To demonstrate non inferiority of a) "FE 999169 Split Dosing Schedule" (one dose on the day before and the second dose on the day of colonoscopy) and b) "FE 999169 Day Before Dosing Schedule" (two doses on the day before colonoscopy) to " Niflec On the Day Dosing Schedule" in subjects requiring colonoscopy.

DETAILED DESCRIPTION:
This was a phase III, randomized, assessor-blinded, parallel-arm, multicenter, study in Japanese patients. Patients, who signed an informed consent and fulfilled all screening criteria, were randomized in a 1:1:1 ratio to one of the following 3 treatment groups: "FE 999169 Split Dosing Schedule", "FE 999169 Day Before Dosing Schedule" and " Niflec On the Day Dosing Schedule" in subjects requiring colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients, age 20 to 80 years inclusive, requiring colonoscopy
* Female patients should be post-menopausal (women ≥45 years with no menstrual period for at least 12 months without an alternative medical cause), or be surgically sterile, or be using medically approved contraception, throughout the trial period.
* Fertile female patients must have a confirmed negative pregnancy test at screening and randomization
* Patients must have had more than or equal to 3 spontaneous bowel movements per week prior to the colonoscopy
* Written informed consent obtained prior to any study-related procedure

Exclusion Criteria:

* Acute surgical abdominal conditions, such as acute intestinal obstruction or intestinal perforation, diverticulitis, appendicitis. If intestinal obstruction and perforation are suspected, perform appropriate diagnostic studies to rule out these conditions
* Active (acute/exacerbation of/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
* Any prior colorectal surgery, excluding appendectomy, haemorrhoid surgery or prior endoscopic procedures
* Colon disease (history of colonic cancer, toxic megacolon, idiopathic pseudo-obstruction, hypomotility syndrome)
* Gastrointestinal disorder (active ulcer, outlet obstruction, retention, gastroparesis, ileus)
* Ascites.
* Upper gastrointestinal surgery (gastric resection, gastric banding, gastric by-pass)
* Uncontrolled angina and/or Myocardial Infarction (MI) within last 3 months, Congestive Heart Failure (CHF), or uncontrolled hypertension
* Renal insufficiency (any of the serum creatinine, or serum potassium value exceeding the upper limits of the normal range at screening) or a history of this event
* Participation in any other clinical trial during the past 3 months
* Any clinically significant laboratory value at screening, including pre-existing electrolyte abnormality, based on clinical history that the investigators feel may affect the study evaluation
* Hypersensitivity to active ingredients
* Subject who cannot suspend the prohibited medications
* Subjects not appropriate to participate in the study as deemed by the investigator

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (4):
- Japan (4):
  - Investigational site, Chiba
  - Investigational site, Kanagawa
  - Investigational site, Kochi
  - Investigational site, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm [1]: FE 999169: One sachet on the day before colonoscopy, and another sachet on the day of colonoscopy
  FE 999169
- Treatment Arm [2]: FE 999169: Two sachets on the day before colonoscopy
  FE 999169
- Treatment Arm [3]: Niflec: One to two pack(s) on the day of colonoscopy
  Niflec
Period: Overall Study
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Started | 214 | 212 | 211
Intention-To-Treat (ITT) Analysis Set | 214 | 212 | 211
Per Protocol (PP) Analysis Set | 212 | 208 | 205
Safety Analysis Set | 213 | 211 | 208
Completed | 213 | 211 | 205
Not Completed | 1 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Not exposed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat Analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec | Total
Number analyzed (Participants) | 214 | 212 | 211 | 637
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (14.0) | 48.3 (14.3) | 48.1 (14.1) | 48.2 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 100 | 95 | 297
  Male | 112 | 112 | 116 | 340
Height [Mean (Standard Deviation); unit: (m)] | 1.64 (0.080) | 1.64 (0.082) | 1.64 (0.084) | 1.64 (0.082)
Weight [Mean (Standard Deviation); unit: (kg)] | 61.9 (11.6) | 63.1 (13.0) | 62.6 (12.5) | 62.5 (12.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m2)] | 22.9 (3.20) | 23.2 (3.59) | 23.2 (3.72) | 23.1 (3.51)

OUTCOME MEASURES:

1. Primary Outcome: The Efficacy Rate Based on the Overall Colon Cleansing Effect as Assessed by the Independent Central Judging Committee Using the Japanese Colon Cleansing Scale
Description: The efficacy rate was based on the overall colon cleansing effect as assessed by the independent central judging committee: the rate of responders who were defined as subjects with a 1 or 2 rating in each colon segment on the Japanese colon cleansing scale, which has scale of 1 (Excellent observation) to 5 (Unable to judge). One of the 5 ratings to each of the colon segments (rectum, sigmoid colon, descending colon, transverse colon, and ascending colon/cecum) was given according to the description and the representative pictures of each rating. A subject who had a 1 or 2 rating in each colon segment was counted as a responder in the overall colon cleansing effect. Otherwise they were counted as a non-responder.
Time Frame: Day 1 (day of colonoscopy)
Population: Intention-To-Treat Analysis set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Number analyzed (Participants) | 214 | 212 | 211
percentage of participants | 97.7 | 92.0 | 95.3

2. Secondary Outcome: The Efficacy Rate Based on the Overall Colon Cleansing Effect Assessed by the Investigators at the Sites Using the Japanese Colon Cleansing Scale
Description: The efficacy rate was based on the overall colon cleansing effect as assessed by the investigators at sites: the rate of responders who were defined as subjects with a 1 or 2 rating in each colon segment on the Japanese colon cleansing scale, which has scale of 1 (Excellent observation) to 5 (Unable to judge). One of the 5 ratings to each of the colon segments (rectum, sigmoid colon, descending colon, transverse colon, and ascending colon/cecum) was given according to the description and the representative pictures of each rating. A subject who had a 1 or 2 rating in each colon segment was counted as a responder in the overall colon cleansing effect. Otherwise they were counted as a non-responder.
Time Frame: Day 1 (day of colonoscopy)
Population: Intention-To-Treat Analysis set
Measure: Number; unit: percentage of participants
Groups:
- Treatment Arm [1]: FE 999169: One sachet of the day before colonoscopy, and another sachet on the day of colonoscopy
  FE 999169
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Number analyzed (Participants) | 214 | 212 | 211
percentage of participants | 88.8 | 79.7 | 93.4

3. Secondary Outcome: The Total Scores of the Colon Cleansing Effect by the Investigators at Sites Using the Ottawa Scale
Description: The total Ottawa scale score was calculated by adding the ratings (0 to 4) for each of the three colon segments, Ascending colon (ascending, cecum), Mid colon (transverse, descending), and Recto-sigmoid colon, in addition to the overall fluid quantity rating (0 (small), 1 (medium), or 2 (large) ). This gave a sum of 0 (best) to 12 (worst) for overall assessment of colon cleansing, and an additional 0 to 2 for the global fluid quantity rating. The final range of the score was from 0 (excellent) to 14 (solid stool in each colon segment and lots of fluid).
Time Frame: Day 1 (day of colonoscopy)
Population: Intention-To-Treat Analysis set
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Number analyzed (Participants) | 214 | 212 | 211
units on a scale | 4.31 [3.94 to 4.67] | 5.18 [4.81 to 5.54] | 2.33 [1.96 to 2.70]

4. Secondary Outcome: Evaluation of Acceptability of the Investigational Medicinal Products (IMPs) by Subjects Using a Questionnaire
Description: The mean score of subjects who gave favourable impression on their assigned IMPs with 3 or 5 points scales, and the frequency of the response for yes/no questions was summarized in each of question for each treatment arm.
  * Ease of consuming the assigned IMPs with a scale of 1(Very easy) to 5 (Very difficult)
  * Overall impression of the assigned IMPs with a scale of 1(Excellent) to 5 (Bad)
  * Taste of the assigned IMPs with a scale of 1 (Excellent) to 5 (Bad)
  * Volume of the assigned IMPs with a scale of 1(Very much) to 3 (No problem)
  * Impression of the assigned IMPs compared with other colon cleansing products with a scale of 1 (Much better) to 5 (Much worse)
Time Frame: Day 0 - Day 1
Population: Intention-To-Treat Analysis set
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Number analyzed (Participants) | 214 | 212 | 211
units on a scale
  IMP compliance, easy or difficult | 1.86 [1.75 to 1.97] | 1.98 [1.87 to 2.08] | 3.08 [2.97 to 3.19]
  Overall impression of assigned IMP | 2.07 [1.97 to 2.18] | 2.10 [2.00 to 2.21] | 2.85 [2.75 to 2.95]
  Taste of assigned IMP | 2.08 [1.96 to 2.19] | 2.23 [2.12 to 2.35] | 3.19 [3.08 to 3.31]
  Volume of IMP consumption | 2.90 [2.84 to 2.97] | 2.89 [2.82 to 2.96] | 2.23 [2.17 to 2.30]
  Comparison with previously colon cleansing | 1.83 [1.52 to 2.14] | 2.22 [1.86 to 2.58] | 2.77 [2.48 to 3.06]

5. Secondary Outcome: Evaluation of Acceptability of the Investigational Medicinal Products (IMPs) by Subjects Using a Questionnaire
Description: The frequency of the response for yes/no questions was summarized in each of question for each treatment arm.
  * Whether or not a subject will request for the assigned IMPs again when the next colonoscopy is needed, with yes-or-no answer
  * Whether or not a subject will refuse the assigned IMPs when it is prescribed for the next colonoscopy, with yes-or-no answer
Time Frame: Day 0 - Day 1
Population: Intention-To-Treat Analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Number analyzed (Participants) | 214 | 212 | 211
percentage of participants
  Wish to use the same drug in future | 92.3 [87.8 to 95.2] | 88.5 [83.4 to 92.1] | 60.9 [54.0 to 67.3]
  Refuse to use the same drug in future | 2.7 [1.2 to 5.8] | 4.5 [2.4 to 8.3] | 11.2 [7.5 to 16.3]

ADVERSE EVENTS:
Arm/Group | Treatment Arm [1]: FE 999169 | Treatment Arm [2]: FE 999169 | Treatment Arm [3]: Niflec
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/211 | 1/208
Other Adverse Events (participants affected / at risk) | 6/213 | 9/211 | 5/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm [1]: FE 999169 (N=213) | Treatment Arm [2]: FE 999169 (N=211) | Treatment Arm [3]: Niflec (N=208)
Post-procedual haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — The Investigator reported the event to be related with the endoscopic mucosal resection procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm [1]: FE 999169 (N=213) | Treatment Arm [2]: FE 999169 (N=211) | Treatment Arm [3]: Niflec (N=208)
Nausea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 5 (5)
Blood magnesium increased (Investigations) | 2 (2) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.